CLINICAL TRIAL: NCT06216626
Title: Assessing the Effects of a Daily Prebiotic Fibre Blend on Inflammation, the Gut Microbiome, and Self-Report Measures of Mental Health in Individuals With Metabolic Syndrome
Brief Title: PRebiotic Intervention for Metabolic and MEntal Health (PRIME)
Acronym: PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myota GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRIME
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome; Anxiety; Mood; Stress
Keywords: gut microbiome; inflammation; mental health
MeSH Terms: conditions — Metabolic Syndrome; Anxiety Disorders; Inflammation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The current protocol is an open-label parallel randomised controlled trial. Participants will be randomised into one of two study arms: a prebiotic fibre intervention arm or control arm (standard of care - Heart UK's Healthy Eating Guidelines).
  Participants in the fibre intervention arm will consume 10g of a powdered fibre mix daily for 12 weeks. Both groups will not receive any additional nutrition support beyond Heart UK Healthy Eating Guidelines during the intervention. Participants will be instructed to maintain their normal lifestyle and diet, and avoid consuming other probiotic or prebiotic (fibre-based) products during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic fibre (Experimental): The treatment group will consume 10g per day of a diverse prebiotic fibre supplement. Supplements are powdered and unflavoured, and given to the participants in 300g packets lasting for 30 days. A 10g scoop is included in each packet and participants are advised to consume one level scoop at any time of the day. Participants are provided with examples on how to consume the supplement (e.g., breakfast cereal, coffee, tea, water).
  Interventions: Dietary Supplement: myota's prebiotic fibre blend
- Control (Active Comparator): Participants are provided with standard of care (dietary advice). Recommendations for diet and lifestyle advice are provided by a UK-registered GP, and follow the Heart UK's Healthy Eating Guidelines. These recommendations emphasise a Mediterranean diet, rich in fruit, vegetables, and healthy fats (omega-3 fatty acids), while reducing refined sugar, salt, processed foods, and alcohol intake. The Mediterranean diet is considered a gold-standard for participants with MetS and poor mental health.
  Interventions: Dietary Supplement: myota's prebiotic fibre blend

INTERVENTIONS:
Dietary Supplement: myota's prebiotic fibre blend — Each 10g daily serve of supplement contains the following fibres:
  * Fructooligosaccharides
  * Inulin
  * Resistant dextrin
  * Resistant maltodextrin
  * Partially hydrolysed guar gum
  * Guar gum

SUMMARY:
The purpose of the study is to determine whether a daily prebiotic fibre blend can reduce systemic inflammation, dyslipidemia, and self-report measures of mental health in individuals with metabolic syndrome. This study will help shape a larger randomised controlled study (RCT) powered to assess efficacy in a bigger cohort of patients.

Primary outcome measures will explore the efficacy of a prebiotic fibre blend on systemic inflammation. Secondary and exploratory outcomes measures will explore the efficacy of the prebiotic blend on clinical biomarkers associated with cardiometabolic risk factors, microbiota features, and mental health. Using these data, we will also estimate in-year savings for the NHS in the metabolic syndrome population on a per participant basis.

DETAILED DESCRIPTION:
Metabolic syndrome is not a chronic disease, but a cluster of metabolic abnormalities including central obesity, insulin resistance, hyperglycemia, hypertension, and dyslipidemia. In the UK, it's estimated that 1 in 3 adults aged 50 years or over meets the criteria of metabolic syndrome. Emerging evidence suggests that metabolic syndrome is associated with low-grade systemic inflammation, which is thought to play a critical role in the subsequent pathogenesis of various metabolic and cardiovascular diseases. In fact, the inflammatory biomarker, high-sensitivity (hs)-CRP, has been shown to be predictive of whether metabolic syndrome progresses to a chronic disease, including cardiovascular disease (CVD), type 2 diabetes (T2D), and cancer mortality. Alongside metabolic disturbances, recent studies have shown that repeated (or long-term) exposure to systemic inflammation is also associated with an increased risk of future depressive and anxiety symptoms, potentially acting via the blood-brain barrier (BBB) interface.

From both a physical and mental health standpoint, it's clear that novel interventions, beyond pharmacotherapy, are needed to reverse the progression of metabolic syndrome, and reduce the risk of developing a long-term chronic disease, and poor mental health.

It is well established that dietary fibre plays a critical role in reducing symptoms of metabolic syndrome, including improvements in insulin sensitivity, glucose metabolism, lipid profile, and blood pressure. Specifically, dietary fibre has been shown to reduce cholesterol levels by binding to bile acids and promoting their excretion, as well as by decreasing the absorption of dietary cholesterol. Additionally, dietary fibre can slow the absorption of carbohydrates and reduce post-prandial glucose spikes, which may contribute to improvements in insulin sensitivity and metabolic health.

Growing evidence also suggests that the mechanisms underlying the benefits of fibre are thought to be mediated, at least in part, by the gut microbiota and their metabolites, such as short-chain fatty acids (SCFAs). A recent systematic review and meta-analysis of 10 randomised controlled trials found that increased intake of dietary fibre was associated with significant improvements in fasting glucose, insulin resistance, total cholesterol, and low-density lipoprotein (LDL) cholesterol levels in individuals with type 2 diabetes. Furthermore, a randomised controlled trial in individuals with metabolic syndrome found that supplementation with a prebiotic fibre blend led to significant reductions in fasting glucose, insulin resistance, and inflammatory markers. Therefore, increasing prebiotic fibre intake may represent a promising strategy for the prevention and management of metabolic symptoms, but remains poorly understood.

Prebiotics are specific types of fibres found in foods like onion, garlic, artichokes, asparagus, leeks, and chicory root. However, to reap the benefits of prebiotics for given health indications, this requires someone to consume roughly 5-10 onions a day. Prebiotic fibre blends (in powder form) are derived from a diversity of plant-based sources, and allows for the study of prebiotic-based benefits in a feasible, easy, measurable, and controlled way.

In this current study, we aim to assess the effects of a daily prebiotic fibre blend on systemic inflammation, the gut microbiome, lipid profiles, and self-report measures of mental health in individuals with metabolic syndrome. The study will be conducted over 12 weeks, and the findings may provide new insights into the potential role of prebiotics in the prevention and management of physical and mental health risk factors associated with chronic disease.

The study population will include adults aged 18-75 years who meet the criteria for metabolic syndrome. To promote the inclusion and diversity of participants across England, this study will be conducted remotely, by posting participants the at-home collection kits (stool and finger prick tests) and online surveys. This gives access to participants who would otherwise not be able to take part in research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-75 years with a diagnosis of Metabolic Syndrome (MetS), yet not receiving treatment for their symptoms
* MetS is diagnosed using the IDF criteria (Alberti, Zimmet & Shaw, 2006). MetS is defined as having abdominal obesity (waist circumference ≥ 94 cm in men, and ≥ 80 cm in women) plus two or more of the following: raised triglycerides (≥1.7 mmol/L); reduced HDL-C (< 1.03 mmol/L in men and < 1.29 mmol/L in women); raised systolic blood pressure (≥ 130 mmHg); raised diastolic blood pressure (≥ 85 mmHg); treatment of previously diagnosed hypertension; raised fasting plasma glucose (≥ 5.6 mmol/L); or previously diagnosed with pre-diabetes.
* Capacity to give informed consent
* Ability to comply with study requirements.

Exclusion Criteria:

* Includes a current diagnosis of Type 1 or 2 diabetes or cardiovascular disease
* receiving medications that lower cholesterol, blood pressure, or blood glucose levels
* pregnancy, lactation, or an intent to become pregnant during the course of the study
* continuous antibiotic use for > 3 days within 1 month prior to enrolment
* continuous use of weight-loss drug for > 1 month before screening
* major change in dietary intake in past month (e.g. excluding whole food groups)
* currently consuming large doses of prebiotic or probiotic supplements
* prior use (< 6 months) of any blood glucose or cholesterol lowering medication
* a significant gastrointestinal (GI) condition affecting absorption including (but not limited to) inflammatory bowel disease; weight loss surgery
* irritable bowel disease
* end stage renal disease
* active cancer, or treatment for any cancer, in last 3 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on C-Reactive Protein levels

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale (42-item) | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on Depression, Anxiety and Stress Scale (42-item) scores. Minimum score = 0, maximum score = 126, where higher scores indicate worse outcomes.
Patient Health Questionnaire (PHQ) | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on Patient Health Questionnaire scores. Minimum score = 1, maximum score = 27, where higher scores indicate worse outcomes.
Perceived Stress Scale (PSS) | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on Perceived Stress Scale scores. Minimum score = 0, maximum score = 40, where higher scores indicate worse outcomes.
Generalised Anxiety Disorder (GAD) Scale | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on Generalised Anxiety Disorder Scale scores. Minimum score = 0, maximum score = 21, where higher scores indicate worse outcomes.
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on Gastrointestinal Symptom Rating Scale scores. Scores are calculated for 5 sub-categories: reflux, pain, constipation, diarrhoea, indigestion, where the minimum score is 1 and maximum score is 21, where higher scores indicate worse outcomes.
Gut Microbiome Profiles | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on gut microbiome profiles
Lipid Profiles | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on lipid profiles
Diastolic blood pressure | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on diastolic blood pressure.
Systolic Blood pressure | Baseline and Week 12
  To compare the effect of Myota's prebiotic fibre blend versus standard of care on systolic blood pressure.

OTHER OUTCOMES:
Dietary fibre intake | Baseline and Week 12
  Assess the difference in dietary fibre intake as a confounding variable.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin V Hall, PhD, Principal Investigator — myota health
Locations (1):
- Myota Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
De-identified participants data may be available to other researchers upon reasonable request.